CLINICAL TRIAL: NCT05591313
Title: Acute Exercise Effect on Neurocognitive Function Among Cognitively Normal Late-Middle-Aged Adults With/Without Generic Risk of Alzheimer's Disease: The Moderation Role of Exercise Volume and Apolipoprotein E Genotype
Brief Title: Acute Exercise on Neurocognitive Function Among Adults With/Without Generic Risk of AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yu-Kai Chang, Proffessor, National Taiwan Normal University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PACNL_EV_ERP_APOE
Record Dates: First submitted 2022-10-12; First posted 2022-10-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease 2 Due to Apoe4 Isoform
Keywords: aerobic exercise; APOE genotype; event-related potential; executive function; exercise prescription
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The present study adopted a counterbalanced design. All participants were instructed to complete four counterbalanced treatments: a) longer duration (LI-40), b) moderate-intensity with 30 min (MI-30), c) high-intensity with shorter duration (HI-16), and d) control treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-intensity with longer duration (40-min) exercise (LI-40) (Experimental): The participants were instructed to complete a volume-matched low-intensity with longer duration (40-min) exercise (LI-40) treatment.
  Interventions: Behavioral: LI-40
- Moderate-intensity with 30 min exercise (MI-30) (Experimental): The participants were instructed to complete a volume-matched moderate-intensity with 30 min exercise (MI-30) treatment.
  Interventions: Behavioral: MI-30
- High-intensity with shorter duration (16-min) exercise (HI-16) (Experimental): The participants were instructed to complete a volume-matched high-intensity with shorter duration (16-min) exercise (HI-16) treatment.
  Interventions: Behavioral: HI-16
- Control treatment (CON) (No Intervention): The participants in the control treatment (CON) were instructed to complete book reading for 30-min.

INTERVENTIONS:
Behavioral: LI-40 — Participants were asked to complete a volume-matched light-intensity exercise for 30-min. The exercise volume was pre-determined based on the energy expenditure (kcal) calculated with 5-min warm-up stage, 20-min main exercise stage (i.e., moderate intensity as 50%-60 % heart rate reserve, HRR), and 5-min cool-down stage.
  Other Names: Light intensity 40-min exercise
  Arms: Low-intensity with longer duration (40-min) exercise (LI-40)
Behavioral: MI-30 — Participants were asked to complete a volume-matched moderate-intensity exercise for 20-min. The exercise volume was pre-determined based on the energy expenditure (kcal) calculated with 5-min warm-up stage, 20-min main exercise stage (i.e., moderate intensity as 50%-60 % heart rate reserve, HRR), and 5-min cool-down stage.
  Other Names: Moderate intensity 30-min exercise
  Arms: Moderate-intensity with 30 min exercise (MI-30)
Behavioral: HI-16 — Participants were asked to complete a volume-matched high-intensity exercise for 16-min. The exercise volume was pre-determined based on the energy expenditure (kcal) calculated with 5-min warm-up stage, 20-min main exercise stage (i.e., moderate intensity as 50%-60 % heart rate reserve, HRR), and 5-min cool-down stage.
  Other Names: High intensity 16-min exercise
  Arms: High-intensity with shorter duration (16-min) exercise (HI-16)

SUMMARY:
This study explores the acute exercise effect on neurocognitive function and also its potential moderators in an exercise setting and Apolipoprotein E (APOE) genetic risk.

DETAILED DESCRIPTION:
Acute exercise has emerged as a modifier to multiple aspects of cognitive function; however, its effect on populations with different risks of Alzheimer's disease (AD) and the role of exercise variance and APOE genotype within the effect reminds underestimated. The current study aimed to examine the acute exercise effect on neurocognitive function from behavioral and neuroelectric perspectives among cognitively normal late-middle-aged adults. Additionally, we determined whether variations in exercise intensity and duration and the presence of the APOE ɛ4 allele modulated the effect.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 50 and 70 years old
2. Normal or corrected-to-normal vision based on the minimal 20/20 standard
3. Cognitively normal as mini-mental state examination scores (MMSE) > 26

Exclusion Criteria:

1. Neurological or psychiatric disorders
2. Cardiovascular disease
3. Risk of cardiovascular fitness assessment based on the Physical Activity Readiness Questionnaire (PAR-Q)
4. Red-green color blindness.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Stroop task: Response time | Participants were required to complete the Stroop task approximately 30 min following the cessation of each acute exercise treatment or the 30-min reading.
  A computerized Stroop task was used to assess participants' inhibitory control and basic information processing. The response time of the correct responses was calculated for the first behavioral index.
Stroop task: Accuracy | Participants were required to complete the Stroop task approximately 30 min following the cessation of each acute exercise treatment or the 30-min reading.
  A computerized Stroop task was used to assess participants' inhibitory control and basic information processing. The accuracy was calculated for the second behavioral index.
Event-related potential: P3 amplitude | Participants were required to complete the Stroop task while EEG activity was continuously recorded approximately 30 min following the cessation of each acute exercise treatment or the 30-min reading.
  The event-related potential from parietal electrodes (i.e., P3, Pz, and P4) were initially outputted for the mean P3 amplitude; the averaged mean P3 amplitudes from parietal electrodes was then calculated as the neuroelectrical indices.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Kai Chang, Ph.D., Study Director — Department of Physical Education and Sport Sciences, National Taiwan Normal University
Locations (1):
- Department of Physical Education and Sport Sciences, National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data are available upon request.

REFERENCES:
- [Derived] Chang YK, Etnier JL, Li RH, Ren FF, Ai JY, Chu CH. Acute Exercise Effect on Neurocognitive Function Among Cognitively Normal Late-Middle-Aged Adults With/Without Genetic Risk of AD: The Moderating Role of Exercise Volume and APOE Genotype. J Gerontol A Biol Sci Med Sci. 2024 Feb 1;79(2):glad179. doi: 10.1093/gerona/glad179. PMID 37526237